CLINICAL TRIAL: NCT07129928
Title: Organizational Strategies and Psychosocial Skills for Maintaining Physical Activity After a Depressive Episode: a 3-month Post-rehabilitation Study.
Acronym: AP&Depression
Status: Not yet recruiting | Type: Observational
Sponsor: Hopital La Musse (Other)
Collaborators: Clinique des portes de l'Eure (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-A00592-47
Record Dates: First submitted 2025-07-02; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Physical Activity; Depression Disorder; Rehabilitation; Organizational Behavior
Keywords: Physical activity; depression; Rehabilitation; Organizational strategies; Psychosocial skills; Determinants of physical activity
MeSH Terms: conditions — Motor Activity; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interview: After recruiting the participants and obtaining their non-opposition to take part in the study, each individual will take part in a semi-structured interview during their 3-month post-stay assessment at the Rehabilitation Center (CDR).

SUMMARY:
With nearly 280 million people affected worldwide (2022), the management of depression represents a major public health issue. The study titled "Organizational Strategies and Psychosocial Skills to Maintain Physical Activity after a Depressive Episode: A 3-Month Post-Rehabilitation Study" (AP&Depression) fits within this context. Physical activity (PA) is now recognized as an effective complementary therapy to pharmacological and psychotherapeutic treatments, helping to regulate mood and reduce depressive symptoms. However, despite these proven benefits, individuals who have experienced a depressive episode often struggle to maintain regular physical activity once they leave the hospital setting. This study aims to identify the mechanisms that influence the continuation of PA after hospitalization by exploring organizational strategies, psychosocial skills, and individual determinants involved in this process.

Depression is a debilitating illness characterized by persistent sadness, loss of interest, chronic fatigue, and impaired cognitive and physical abilities (DSM-5, 2013). Among the aggravating factors, sedentary behavior plays a key role, whereas PA is associated with a significant reduction in the risk of relapse. Yet, 67.8% of individuals with depression do not meet the recommended 150 minutes of weekly PA, and this figure rises to 85.7% when activity is measured objectively. This situation is explained by several barriers: lack of motivation, low self-efficacy, fluctuating mood disorders, social isolation, and limited access to exercise facilities. Conversely, certain factors facilitate the resumption of PA after a depressive episode, including structured support, the establishment of routines, social support, and therapeutic education.

The study relies on a qualitative methodology using semi-structured interviews conducted with 15 patients who stayed at the Rehabilitation Center of the Clinique des Portes de l'Eure. Participants are selected according to the following criteria: aged over 18, medically diagnosed with a depressive episode, underwent rehabilitation, and completed an initial assessment at the Maison Sport Santé. They will be interviewed three months after discharge to explore their PA practices. Data will be analyzed using NVivo software, following the COREQ (Consolidated Criteria for Reporting Qualitative Research) guidelines. The analysis of transcripts will help identify the organizational strategies implemented, the psychosocial skills involved, and the individual determinants influencing the maintenance of regular PA.

The expected results should highlight that patients adopt various strategies to maintain PA after hospitalization. Session planning, the gradual integration of PA into daily life, and the anticipation of obstacles are major levers for establishing a sustainable routine. In addition, psychosocial skills, such as stress management and interaction with a support network, emerge as essential elements for maintaining regular physical activity. However, several obstacles may be identified, including persistent fatigue, mood fluctuations, lack of organization, and social isolation. These findings underscore the importance of personalized support after rehabilitation, particularly through mechanisms such as Patient Therapeutic Education (PTE) or individualized follow-up in Maisons Sport Santé.

The aim of this study is to shed light on the mechanisms that enable individuals who have experienced a depressive episode to autonomously maintain physical activity after hospitalization. This research seeks to provide concrete recommendations for improving support during and after hospitalization to enhance adherence to PA. The study's conclusions could contribute to the development of new therapeutic approaches aimed at improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* French-speaking patient
* Patient with a depressive episode diagnosed by a physician
* Patient who completed a stay at the Rehabilitation Center (CDR) at the Clinique des Portes de l'Eure
* Patient at 3 months post-rehabilitation stay
* Patient who completed an initial assessment (T0) at the Maison Sport Santé during the clinic stay

Exclusion Criteria:

* Exacerbation of the condition
* Patient who has already completed a 3-month follow-up assessment at the Maison Sport Santé (MSS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The chosen study population consists of patients who have experienced a depressive episode
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of patients' organizational strategies observed during the semi-structured interview | Day 1
  The primary outcome of this study is the identification of organizational strategies used by patients who have experienced a depressive episode to maintain autonomous physical activity three months after their hospitalization. The objective is to evaluate the mechanisms that support the continuation of physical activity outside the hospital setting and to understand the main driving factors. These strategies will be observed during the semi-structured interview (verbatims analysis).
Identification of patients' psychosocial skills observed during the semi-structured interview | Day 1
  The primary outcome of this study is the identification of psychosocial skills used by patients who have experienced a depressive episode to maintain autonomous physical activity three months after their hospitalization. The objective is to evaluate the mechanisms that support the continuation of physical activity outside the hospital setting and to understand the main driving factors. These skills will be observed during the semi-structured interview (verbatims analysis).
Identification of patients' individual determinants observed during semi-structured interview | Day 1
  The primary outcome of this study is the identification of individual determinants used by patients who have experienced a depressive episode to maintain autonomous physical activity three months after their hospitalization. The objective is to evaluate the mechanisms that support the continuation of physical activity outside the hospital setting and to understand the main driving factors. These determinants will be observed during semi-structured interview (verbatims analysis).

SECONDARY OUTCOMES:
Analyze the specific barriers encountered by these patients in maintaining regular physical activity, through the analysis of semi-structured interviews. | Day 1
  The secondary outcomes focus on analyzing the specific barriers encountered by these patients in maintaining regular physical activity.
  In addition, the study aims to assess the frequency and persistence of physical activity after a stay in the Rehabilitation Center (CDR), by identifying both the obstacles and the facilitators to achieving long-term autonomy in physical activity (analysis of verbatim transcripts following semi-structured interviews).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Musse, Saint-Sébastien-de-Morsent, France

IPD SHARING:
Plan to Share IPD: Undecided